CLINICAL TRIAL: NCT00561184
Title: A Phase II, Open-label, Multi-Center Study to Evaluate Safety and Immunogenicity of a Booster Dose of -H5N1 (Surface Antigen Adjuvanted With MF59C.1) Influenza Vaccine in Non-elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of a Booster Dose of -H5N1 Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V87P1E1; 2007-000165-38
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-02

CONDITIONS: Avian Influenza
Keywords: H5N1 Pandemic
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: H5N1 influenza vaccine
- 2 (Experimental)
  Interventions: Biological: H5N1 influenza vaccine

INTERVENTIONS:
Biological: H5N1 influenza vaccine — One 0.5 ml booster injection 12 months after the second injection, of influenza vaccine containing 7.5 micrograms of H5N1 influenza antigen
  Arms: 1
Biological: H5N1 influenza vaccine — One 0.5 ml booster injection 12 months after the second injection, of influenza vaccine containing 15.0 micrograms of H5N1 influenza antigen
  Arms: 2

SUMMARY:
To assess persistence of antibody titers 17-18 months after primary immunization with two 0.5mL intramuscular (IM) doses of H5N1 influenza vaccine containing H5N1 influenza antigen, as measured by Hemagglutination Inhibition (HI), Single Radial Hemolysis (SRH), and Microneutralization (MN) test

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who previously participated in study V87P1, but did not receive the booster dose on day 202

Exclusion Criteria:

* Pregnant or breastfeeding
* Receipt of another vaccine or any investigational agent within the past 4 weeks
* Surgery planned during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with at least one local reaction between 1 and 7 days after vaccination. | 7 days
Number and percentage of subjects with at least one systemic reaction between 1 and 7 days after vaccination. | 7 days

SECONDARY OUTCOMES:
Number and percentage of subjects with at least one adverse event between day of vaccination and the study termination visit.Safety will be assessed in accordance with available safety data on influenza vaccines. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- Italy (3):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G. D'Annunzio, Via dei Vestini, Chieti
  - 01: Dipartimento di Scienze della Salute, Sezione Igiene e Medicina Preventiva, Università di Genova, Genova
  - 03: Ufficio di Igiene e Sanità Pubblica di Lanciano, ASL Lanciano -Vasto, Via Spaventa, 37,, Lanciano

REFERENCES:
- [Result] Fragapane E, Gasparini R, Schioppa F, Laghi-Pasini F, Montomoli E, Banzhoff A. A heterologous MF59-adjuvanted H5N1 prepandemic influenza booster vaccine induces a robust, cross-reactive immune response in adults and the elderly. Clin Vaccine Immunol. 2010 Nov;17(11):1817-9. doi: 10.1128/CVI.00461-09. Epub 2010 Sep 1. PMID 20810680